CLINICAL TRIAL: NCT00239005
Title: A Study of the Effect of Conversion to Enteric-Coated Mycophenolate Sodium (EC-MPS) on Quality of Life in Patients With Gastrointestinal (GI) Symptoms Related to Mycophenolate Mofetil Therapy After Kidney Transplantation (MYQOL)
Brief Title: Enteric-Coated Mycophenolate Sodium on Quality of Life in Patients With Gastrointestinal Symptoms Related to Mycophenolate Mofetil Therapy After Kidney Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CERL080AGB03; 2004-005071-42
Record Dates: First submitted 2005-10-12; First posted 2005-10-14 (Estimated); Results first posted 2011-03-24 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-02

CONDITIONS: Renal Transplant
Keywords: QoL; GI Side Effects; MPA
MeSH Terms: interventions — Mycophenolic Acid

ARMS (2):
- Mycophenolate Mofetil (MMF) (Active Comparator): 250 mg capsules or 500 mg tablets of mycophenolate mofetil. Daily dose decided by physician, was taken morning and evening.
  Interventions: Drug: Mycophenolate Mofetil (MMF)
- Enteric-Coated Mycophenolate Sodium (EC-MPS ) (Experimental): Oral film-coated gastroresistant tablets containing 360mg or 180mg of mycophenolate sodium. Daily dose decided by the physician, was taken morning and evening.
  Interventions: Drug: Enteric-Coated Mycophenolate Sodium (EC-MPS)

INTERVENTIONS:
Drug: Enteric-Coated Mycophenolate Sodium (EC-MPS)
  Other Names: Myfortic®
  Arms: Enteric-Coated Mycophenolate Sodium (EC-MPS )
Drug: Mycophenolate Mofetil (MMF)
  Other Names: Cellcept®
  Arms: Mycophenolate Mofetil (MMF)

SUMMARY:
This open, multi-center randomized controlled study is designed to investigate the quality of life in patients with mycophenolate mofetil (MMF)-induced gastrointestinal (GI) adverse events after converting to enteric-coated mycophenolate sodium (EC-MPS).

ELIGIBILITY:
Inclusion Criteria:

1. Received kidney transplant
2. Receiving immunosuppressive regimen that includes MMF
3. Patients with GI side effects on standard MMF doses or patients on reduced dose MMF with existing but tolerated/controlled GI side effects.
4. At least 18 years of age
5. Willing to provide written informed consent
6. Able to meet all study requirements including completing questionnaires and completing four study visits.

Exclusion Criteria:

1. Patients with GI symptoms assumed or known not to be caused by medroxyprogesterone acetate (MPA) therapy (e.g. oral bisphosphonate induced, infectious diarrhea)
2. Acute rejection < 1 week prior to study enrollment
3. Woman of child-bearing potential who is planning to become pregnant or is pregnant and/or lactating and who is unwilling to use effective means of contraception
4. Presence of psychiatric illness (i.e., schizophrenia, major depression) that, in the opinion of the site investigator, would interfere with study requirements
5. Undergoing acute medical intervention or hospitalization
6. Any other medical condition that, in the opinion of the site investigator based on recall or chart review, would interfere with completing the study, including, but not limited to, visual problems or cognitive impairment.
7. Receiving any investigational drug or have received any investigational drug within 30 days prior to study enrollment.

Additional protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2005-09; Primary Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Magdi Shehata, MBBCh, MD, FRCS, Principal Investigator — Director of Transplantation, Nottingham City Hospital, Nottingham
Locations (1):
- Novartis Investigative Site, Nottingham, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In total, 135 patients were screened. One patient was not randomized due to an SAE prior to the randomization visit. Out of 134 randomized patients, 5 withdrew before taking study drug. Analysis population: 68 in EC-MPS, 61 in MMF.
Groups:
- Enteric-Coated Mycophenolate Sodium (EC-MPS): Oral film-coated gastroresistant tablets containing 360mg or 180mg of mycophenolate sodium. Daily dose decided by the physician, was taken morning and evening.
Period: Overall Study
Arm/Group | Enteric-Coated Mycophenolate Sodium (EC-MPS) | Mycophenolate Mofetil (MMF)
Started | 69 | 65
Intention-to-treat Population (ITT) | 68 | 61
Completed | 57 | 53
Not Completed | 12 | 12
Not completed — Adverse Event | 6 | 6
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Unsatisfactory Therapeutic effect | 2 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Subj. cond. no longer needs study drug | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enteric-Coated Mycophenolate Sodium (EC-MPS) | Mycophenolate Mofetil (MMF) | Total
Number analyzed (Participants) | 68 | 61 | 129
Age, Customized [Number; unit: participants] — Baseline Measures are based on Intention to treat (ITT) population.
  participants
    <65 years | 65 | 51 | 116
    >=65 years | 3 | 10 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 25 | 56
  Male | 37 | 36 | 73

OUTCOME MEASURES:

1. Primary Outcome: Mycophenolic Acid (MPA) Maintenance Treatment
Description: The primary assessment was based on the percentage of patients who were maintained at week 13 on a dose at least one dose equivalent greater than at baseline (visit 2/week 1). A dose equivalent was defined as EC-MPS 180 mg/day or MMF 250 mg/day.
Time Frame: at week 13 (last visit)
Population: The intent-to-treat (ITT) population consisted of all randomized patients who provided baseline and at least 1 post-baseline assessment of the primary variable.
Measure: Number (95% Confidence Interval); unit: Percentage of Patients
Arm/Group | Enteric-Coated Mycophenolate Sodium (EC-MPS) | Mycophenolate Mofetil (MMF)
Number analyzed (Participants) | 68 | 61
Percentage of Patients | 47.06 [34.83 to 59.55] | 16.39 [8.15 to 28.09]

2. Secondary Outcome: Changes in Gastrointestinal (GI) Symptoms as Measured by the Gastrointestinal Symptom Rating Scale (GSRS).
Description: The GSRS is a 15-item instrument designed to assess the impact of upper and lower GI symptoms. There are five subscales: reflux, diarrhea, constipation, abdominal pain, and indigestion-each of which produces a mean subscale score ranging from 1 (no discomfort) to 7 (very severe discomfort). A higher score represents greater impairment of quality of life due to GI symptoms (range from 1 to 7).
Time Frame: At week 3 and week 13 (last visit)
Population: Intention to treat (ITT) population consisted of all randomized patients who provided baseline and at least 1 post-baseline assessment of the primary variable. In this analysis patients who completed GSRS questionnaire in visit 2 (week 1), visit 3 (week 3) and visit 4 (week 13) were included.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Enteric-Coated Mycophenolate Sodium (EC-MPS) | Mycophenolate Mofetil (MMF)
Number analyzed (Participants) | 61 | 59
Units on a scale
  Week 3: change in GSRS Total Score (N= 61, 59) | -0.63 (0.139) | -0.32 (0.142)
  Week 13: change in GSRS Total Score (N= 60, 56) | -0.44 (0.165) | -0.25 (0.169)

3. Secondary Outcome: Changes in Gastrointestinal Symptoms as Measured by the Gastrointestinal Quality of Life Index (GIQLI).
Description: Health-related quality of life (HRQoL)was assessed by the Gastrointestinal Quality of Life Index (GIQLI). The GIQLI is a 36-item questionnaire to assess the impact of GI disease on daily life. The GIQLI also has five different subscales (GI symptoms, emotional status, physical and social functions, and stress of medical treatment) producing a total score of the 36 items. Lower scores represent more dysfunction. A higher score represents a better quality of life (range from 0 to 144).
Time Frame: At week 3 and week 13 (last visit)
Population: Intention to treat (ITT) population consisted of all randomized patients who provided baseline and at least 1 post-baseline assessment of the primary variable. In this analysis patients who completed GIQLI questionnaire in visit 2 (week 1), visit 3 (week 3) and visit 4 (week 13) were included.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Enteric-Coated Mycophenolate Sodium (EC-MPS) | Mycophenolate Mofetil (MMF)
Number analyzed (Participants) | 61 | 58
Units on a scale
  Week 3: change in GIQLI Total Score (N= 61, 58) | 11.65 (3.470) | 6.08 (3.549)
  Week 13: change in GIQLI Total Score (N= 60, 56) | 4.84 (4.331) | 1.77 (4.458)

ADVERSE EVENTS:
Time Frame: 13 weeks
Description: The Safety population consisted of all randomized patients who had at least one post-baseline safety assessment.
Arm/Group | Enteric-Coated Mycophenolate Sodium (EC-MPS) | Mycophenolate Mofetil (MMF)
Serious Adverse Events (participants affected / at risk) | 9/68 | 7/61
Other Adverse Events (participants affected / at risk) | 25/68 | 26/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enteric-Coated Mycophenolate Sodium (EC-MPS) (N=68) | Mycophenolate Mofetil (MMF) (N=61)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Chills (General disorders) | 0 | 1
Pyrexia (General disorders) | 3 | 0
Cytomegalovirus infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 2 | 1
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aortic dissection (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Enteric-Coated Mycophenolate Sodium (EC-MPS) (N=68) | Mycophenolate Mofetil (MMF) (N=61)
Abdominal pain (Gastrointestinal disorders) | 4 | 1
Diarrhoea (Gastrointestinal disorders) | 12 | 12
Dyspepsia (Gastrointestinal disorders) | 3 | 5
Nausea (Gastrointestinal disorders) | 3 | 4
Vomiting (Gastrointestinal disorders) | 5 | 4
Lower respiratory tract infection (Infections and infestations) | 2 | 4
Nasopharyngitis (Infections and infestations) | 4 | 4
Urinary tract infection (Infections and infestations) | 2 | 4
Headache (Nervous system disorders) | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.